CLINICAL TRIAL: NCT04691115
Title: AM1476 - A Phase I, Double-blind, Placebo-controlled, Single- and Multiple-oral Dose, Safety, Tolerability, and Pharmacokinetic Study in Healthy Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of AM1476 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AnaMar AB (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1476-291-001
Record Dates: First submitted 2020-12-15; First posted 2020-12-31 (Actual); Results first posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-02

CONDITIONS: Safety; Tolerability

STUDY DESIGN:
Intervention Model Description: Part A (SAD) Within each group, subjects will be randomised in a 3:1 ratio to receive either AM1476 (n=6) or placebo (n=2). The first 2 subjects in each group will be dosed in a sentinel fashion; 1 subject will receive AM1476 and the other will receive placebo as randomised.
  Part B (MAD) Within each group, subjects will be randomised in a 3:1 ratio to receive either AM1476 (n=6) or placebo (n=2).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Part A, Group 1: AM1476 1 mg (Experimental): Part A, Group 1: AM1476 1 mg capsule, orally once on Day 1 in fasted state
  Interventions: Drug: AM1476
- Part A, Group 2: AM1476 5 mg (Experimental): Part A, Group 2: AM1476 5 mg capsule, orally once on Days 1 in fasted state
  Interventions: Drug: AM1476
- Part A, Group 3: AM1476 25 mg (Experimental): Part A, Group 3: AM1476 25 mg capsule, orally once on Days 1 in fasted state
  Interventions: Drug: AM1476
- Part A, Group 4: AM1476 125 mg (Experimental): Part A, Group 4: AM1476 125 mg capsule, orally once on Days 1 in fasted state
  Interventions: Drug: AM1476
- Part A, Group 5: AM1476 375 mg (Experimental): Part A, Group 5: AM1476 375 mg capsule, orally once on Days 1 in fasted state
  Interventions: Drug: AM1476
- Part A, Group 6: AM1476 650 mg (Experimental): Part A, Group 6: AM1476 650 mg capsule, orally once on Days 1 in fasted state
  Interventions: Drug: AM1476
- Part A, Group 7: AM1476 950 mg (Experimental): Part A, Group 7: AM1476 950 mg capsule, orally once on Days 1 in fasted state
  Interventions: Drug: AM1476
- Part A, Group 8: AM1476 1500 mg (Experimental): Part A, Group 8: AM1476 1500 mg capsule, orally once on Days 1 in fasted state
  Interventions: Drug: AM1476
- Part A, Group 9: AM1476 2400 mg (Experimental): Part A, Group 9: AM1476 2400 mg capsule, orally once on Days 1 in fasted state
  Interventions: Drug: AM1476
- Part A, Groups 1 to 9: Placebo (Placebo Comparator): Part A, Groups 1 to 9: AM1476 placebo-matching capsule, orally once on Days 1 in fasted state
  Interventions: Drug: Placebo
- Part B, Group 1: AM1476 100 mg QD (once daily) (Experimental): Part B, Group 1: AM1476 100 mg capsule, orally once on Days 1-10 in fasted state
  Interventions: Drug: AM1476
- Part B, Group 2: AM1476 375 mg BID (twice daily) (Experimental): Part B, Group 2: AM1476 375 mg capsule, orally twice on Days 1-9 and once on Days 10 in fasted state
  Interventions: Drug: AM1476
- Part B, Group 3: AM1476 500 mg BID (Experimental): Part B, Group 3: AM1476 500 mg capsule, orally twice on Days 1-9 and once on Days 10 in fasted state
  Interventions: Drug: AM1476
- Part B, Groups 1 to 3: Placebo (Placebo Comparator): Part B, Groups 1 to 3: AM1476 placebo-matching capsule, orally once or twice on Days 1-10 in fasted state
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AM1476 — AM1476 Capsules
  Arms: Part A, Group 1: AM1476 1 mg; Part A, Group 2: AM1476 5 mg; Part A, Group 3: AM1476 25 mg; Part A, Group 4: AM1476 125 mg; Part A, Group 5: AM1476 375 mg; Part A, Group 6: AM1476 650 mg; Part A, Group 7: AM1476 950 mg; Part A, Group 8: AM1476 1500 mg; Part A, Group 9: AM1476 2400 mg; Part B, Group 1: AM1476 100 mg QD (once daily); Part B, Group 2: AM1476 375 mg BID (twice daily); Part B, Group 3: AM1476 500 mg BID
Drug: Placebo — Placebo Capsules
  Arms: Part A, Groups 1 to 9: Placebo; Part B, Groups 1 to 3: Placebo

SUMMARY:
This is a First in Human (FIH), double-blind, randomised, placebo-controlled study designed to evaluate safety, tolerability and pharmacokinetics (PK) of single and multiple ascending oral doses of AM1476 in healthy subjects.

DETAILED DESCRIPTION:
Part A (SAD); In the SAD part of the study, single oral doses of AM1476 will be administered in up to 9 sequential groups, each consisting of 8 subjects randomised to receive either AM1476 or placebo in a 3:1 ratio. The first 2 subjects in each group will be dosed in a sentinel fashion, 1 subject will receive AM1476 and the other will receive placebo as randomised.

Part B (MAD); The MAD part of the study will explore multiple ascending dosing of AM1476 for 10 days. AM1476 will be administered in up to 6 sequential groups, each consisting of 8 subjects randomised to receive either AM1476 or placebo in a 3:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any race, between 18 and 60 years of age, inclusive.
2. A body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive.
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital non-haemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at Screening and/or Check-in (Day -1) as assessed by the Investigator (or designee).
4. Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception as detailed in Appendix 4.
5. Able to comprehend and willing to sign an ICF and to abide by the study restrictions.

Exclusion Criteria

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
3. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).
4. Any of the following observed in at least 2 of 3 ECG measurements performed:

   1. QTcF > 450 msec.
   2. QRS duration > 110 msec.
   3. PR interval > 220 msec.
   4. findings which would make QTc measurements difficult or QTc data uninterpretable.
5. Any history of additional risk factors for torsades de pointes (eg, heart failure, hypokalaemia, family history of long QT syndrome).
6. Any history or current controlled or uncontrolled hypertension or systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg confirmed by repeat measurement.
7. History of alcoholism or drug/chemical abuse within 2 years prior to Check-in (Day -1).
8. Alcohol consumption of > 21 units per week for males and > 14 units per week for females. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
9. Positive alcohol breath test result or positive urine drug screen (confirmed by repeat) at Screening or Check-in (Day -1).
10. Positive hepatitis panel and/or positive human immunodeficiency virus test (Appendix 2).
11. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 90 days prior to dosing.
12. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's Wort, within 30 days prior to dosing, unless deemed acceptable by the Investigator (or designee).
13. Use or intend to use any prescription medications/products other than hormone replacement therapy, oral, implantable, transdermal, injectable, or intrauterine contraceptives within 14 days prior to dosing, unless deemed acceptable by the Investigator (or designee).
14. Use or intend to use slow release medications/products considered to still be active within 14 days prior to Check-in (Day -1), unless deemed acceptable by the Investigator (or designee).
15. Use or intend to use any non-prescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 7 days prior to Check-in (Day -1), unless deemed acceptable by the Investigator (or designee).
16. Use of tobacco- or nicotine-containing products within 3 months prior to Check-in (Day -1) or positive cotinine at Screening or Check-in (Day -1).
17. Ingestion of poppy seeds, Seville orange, or grapefruit-containing foods or beverages within 7 days prior to Check-in (Day -1).
18. Subjects who are vegetarians, vegans, or are unable to consume the high-fat breakfast (subjects who will participate in a food-effect evaluation only).
19. Receipt of blood products within 2 months prior to Check-in (Day -1).
20. Donation of blood from 3 months prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.
21. Poor peripheral venous access.
22. Have previously completed or withdrawn from this study or any other study investigating AM1476, and have previously received AM1476.
23. Subjects who are not willing to minimise or avoid exposure to natural or artificial sunlight (tanning beds or UVA/B treatment) following administration of study drug until 2 weeks after the last dose.
24. Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part B, Group 1: AM1476 100 mg QD: Part B, Group 1: AM1476 100 mg capsule, orally once on Days 1-10 in fasted state
  AM1476: AM1476 Capsules
- Part B, Group 2: AM1476 375 mg BID: Part B, Group 2: AM1476 375 mg capsule, orally twice on Days 1-9 and once on Days 10 in fasted state
  AM1476: AM1476 Capsules
Period: Overall Study
Arm/Group | Part A, Groups 1 to 9: Placebo | Part A, Group 1: AM1476 1 mg | Part A, Group 2: AM1476 5 mg | Part A, Group 3: AM1476 25 mg | Part A, Group 4: AM1476 125 mg | Part A, Group 5: AM1476 375 mg | Part A, Group 6: AM1476 650 mg | Part A, Group 7: AM1476 950 mg | Part A, Group 8: AM1476 1500 mg | Part A, Group 9: AM1476 2400 mg | Part B, Groups 1 to 3: Placebo | Part B, Group 1: AM1476 100 mg QD | Part B, Group 2: AM1476 375 mg BID | Part B, Group 3: AM1476 500 mg BID
Started | 18 | 6 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A, Groups 1 to 9: Placebo | Part A, Group 1: AM1476 1 mg | Part A, Group 2: AM1476 5 mg | Part A, Group 3: AM1476 25 mg | Part A, Group 4: AM1476 125 mg | Part A, Group 5: AM1476 375 mg | Part A, Group 6: AM1476 650 mg | Part A, Group 7: AM1476 950 mg | Part A, Group 8: AM1476 1500 mg | Part A, Group 9: AM1476 2400 mg | Part B, Groups 1 to 3: Placebo | Part B, Group 1: AM1476 100 mg QD | Part B, Group 2: AM1476 375 mg BID | Part B, Group 3: AM1476 500 mg BID | Total
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (12.95) | 42.3 (14.56) | 38.8 (16.63) | 37.0 (14.82) | 38.2 (11.65) | 28.4 (6.21) | 50.8 (11.02) | 37.0 (13.11) | 35.2 (13.99) | 38.5 (15.87) | 37.3 (15.17) | 30.7 (8.19) | 34.3 (14.24) | 28.2 (4.17) | 37.5 (13.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 3 | 3 | 2 | 4 | 3 | 4 | 2 | 1 | 2 | 3 | 2 | 0 | 34
  Male | 14 | 5 | 3 | 3 | 4 | 3 | 3 | 2 | 4 | 5 | 4 | 3 | 4 | 6 | 63
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 18 | 6 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 97
Height [Mean (Standard Deviation); unit: cm] | 174.3 (6.73) | 179.2 (10.38) | 171.0 (9.61) | 176.9 (4.48) | 173.3 (10.25) | 173.3 (9.60) | 173.7 (8.41) | 169.3 (8.87) | 174.2 (5.98) | 181.3 (8.64) | 175.8 (9.41) | 170.8 (8.16) | 174.3 (9.89) | 178.3 (5.35) | 174.6 (8.25)
Body Weight [Mean (Standard Deviation); unit: kg] | 76.91 (13.376) | 85.70 (19.447) | 75.58 (10.193) | 81.35 (11.542) | 78.12 (14.972) | 74.60 (14.594) | 79.93 (10.994) | 76.13 (13.650) | 82.35 (15.599) | 80.93 (14.020) | 81.63 (19.397) | 73.05 (14.729) | 70.98 (15.157) | 78.65 (13.827) | 78.07 (13.925)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 25.23 (3.626) | 26.33 (3.912) | 26.03 (4.479) | 25.98 (3.378) | 25.78 (2.662) | 24.67 (3.119) | 26.45 (2.402) | 26.37 (2.382) | 27.18 (5.115) | 24.55 (3.462) | 26.18 (4.659) | 24.83 (3.435) | 23.15 (2.673) | 24.60 (3.200) | 25.48 (3.451)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: A treatment-emergent adverse-event (TEAE) was defined as an adverse event that started during or after first dosing, or started prior to first dosing and increased in severity after first dosing.
Time Frame: Through study completion, an average of 7 weeks
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Groups 1 to 9: Placebo | Part A, Group 1: AM1476 1 mg | Part A, Group 2: AM1476 5 mg | Part A, Group 3: AM1476 25 mg | Part A, Group 4: AM1476 125 mg | Part A, Group 5: AM1476 375 mg | Part A, Group 6: AM1476 650 mg | Part A, Group 7: AM1476 950 mg | Part A, Group 8: AM1476 1500 mg | Part A, Group 9: AM1476 2400 mg | Part B, Groups 1 to 3: Placebo | Part B, Group 1: AM1476 100 mg QD | Part B, Group 2: AM1476 375 mg BID | Part B, Group 3: AM1476 500 mg BID
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 3 | 0 | 0 | 4 | 1 | 2 | 3 | 2 | 4 | 5 | 6 | 3 | 2 | 4

2. Secondary Outcome: Cmax
Description: maximum plasma concentration
Time Frame: From pre-dose to up to 48 hours post-dose
Population: The pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of AM1476. At the 1 mg AM1476 dose level, the AM1476 concentrations for one participant were below the level of quantification at all timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A, Group 1: AM1476 1 mg | Part A, Group 2: AM1476 5 mg | Part A, Group 3: AM1476 25 mg | Part A, Group 4: AM1476 125 mg | Part A, Group 5: AM1476 375 mg | Part A, Group 6: AM1476 650 mg | Part A, Group 7: AM1476 950 mg | Part A, Group 8: AM1476 1500 mg | Part A, Group 9: AM1476 2400 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6
ng/mL | 0.165 (46.8) | 0.785 (43.4) | 3.83 (36.2) | 30.0 (57.6) | 119 (48.9) | 260 (102.2) | 334 (64.4) | 654 (89.7) | 1250 (35.8)

3. Secondary Outcome: Cmax
Description: maximum plasma concentration
Time Frame: Day 1: From pre-dose up to 24 hours post first dose after QD dosing and from pre-dose up to 12 hours post first dose after BID dosing. Day 10: From pre-dose up to 48 hours post last dose.
Population: The pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of AM1476
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B, Group 1: AM1476 100 mg QD | Part B, Group 2: AM1476 375 mg BID | Part B, Group 3: AM1476 500 mg BID
Number analyzed (Participants) | 6 | 6 | 6
ng/mL
  Day 1 | 18.8 (63.5) | 116 (52.1) | 252 (41.6)
  Day 10 | 26.0 (40.9) | 202 (48.4) | 278 (32.6)

4. Secondary Outcome: Tmax
Description: time to Cmax
Time Frame: From pre-dose to up to 48 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Part A, Group 1: AM1476 1 mg | Part A, Group 2: AM1476 5 mg | Part A, Group 3: AM1476 25 mg | Part A, Group 4: AM1476 125 mg | Part A, Group 5: AM1476 375 mg | Part A, Group 6: AM1476 650 mg | Part A, Group 7: AM1476 950 mg | Part A, Group 8: AM1476 1500 mg | Part A, Group 9: AM1476 2400 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6
hour | 1.50 [0.500 to 3.00] | 1.75 [1.00 to 2.00] | 1.00 [0.500 to 1.00] | 0.983 [0.500 to 1.50] | 1.00 [0.500 to 1.50] | 1.01 [1.00 to 2.00] | 1.51 [1.00 to 2.00] | 1.00 [1.00 to 3.00] | 1.00 [0.500 to 2.00]

5. Secondary Outcome: Tmax
Description: time to Cmax
Time Frame: as for outcome 3
Population: The pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of AM1476
Measure: Median (Full Range); unit: hour
Arm/Group | Part B, Group 1: AM1476 100 mg QD | Part B, Group 2: AM1476 375 mg BID | Part B, Group 3: AM1476 500 mg BID
Number analyzed (Participants) | 6 | 6 | 6
hour
  Day 1 | 0.500 [0.500 to 1.00] | 1.00 [0.500 to 2.00] | 1.00 [0.517 to 1.50]
  Day 10 | 0.775 [0.500 to 2.00] | 1.00 [0.500 to 1.50] | 1.25 [1.00 to 1.50]

6. Secondary Outcome: T½
Description: terminal half-life
Time Frame: From pre-dose to up to 48 hours post-dose
Population: The pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of AM1476. At the 1 mg AM1476 dose level, the t½ was not calculable due to the limited quantifiable AM1476 concentrations available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Part A, Group 1: AM1476 1 mg | Part A, Group 2: AM1476 5 mg | Part A, Group 3: AM1476 25 mg | Part A, Group 4: AM1476 125 mg | Part A, Group 5: AM1476 375 mg | Part A, Group 6: AM1476 650 mg | Part A, Group 7: AM1476 950 mg | Part A, Group 8: AM1476 1500 mg | Part A, Group 9: AM1476 2400 mg
Number analyzed (Participants) | 0 | 5 | 6 | 6 | 6 | 6 | 5 | 6 | 6
hour |  | 2.52 (14.8) | 4.58 (49.4) | 8.34 (40.6) | 13.7 (112.8) | 10.1 (19.5) | 7.84 (9.1) | 8.91 (8.7) | 7.36 (24.1)

7. Secondary Outcome: T½
Description: terminal half-life
Time Frame: as for outcome 3
Population: The pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of AM1476.
  A reliable characterization of the terminal half-life could not be obtained according the calculation criteria in the Statistical analytical plan for 2 participants dosed with 100 mg QD and 1 participant dosed with 375 mg BID on Day 10.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Part B, Group 1: AM1476 100 mg QD | Part B, Group 2: AM1476 375 mg BID | Part B, Group 3: AM1476 500 mg BID
Number analyzed (Participants) | 6 | 6 | 6
hour
  Day 1 | 5.70 (19.6) | 3.23 (8.4) | 2.89 (12.2)
  Day 10: number analyzed (Participants) | 4 | 5 | 6
  Day 10 | 11.4 (27.9) | 12.8 (16.6) | 15.8 (21.6)

8. Secondary Outcome: AUC0-tlast
Description: area under the curve from time 0 to time of the last quantifiable concentration
Time Frame: From pre-dose to up to 48 hours post-dose
Population: The pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of AM1476. At the 1 mg AM1476 dose level, the AUC was not reported for 4 participants due to less than 3 consecutive quantifiable concentrations (calculation criteria in the Statistical analytical plan).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A, Group 1: AM1476 1 mg | Part A, Group 2: AM1476 5 mg | Part A, Group 3: AM1476 25 mg | Part A, Group 4: AM1476 125 mg | Part A, Group 5: AM1476 375 mg | Part A, Group 6: AM1476 650 mg | Part A, Group 7: AM1476 950 mg | Part A, Group 8: AM1476 1500 mg | Part A, Group 9: AM1476 2400 mg
Number analyzed (Participants) | 2 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6
h*ng/mL | NA (NA) — Not calculated as only results from 2 participants | 2.77 (26.1) | 15.0 (26.1) | 113 (33.6) | 312 (44.8) | 882 (73.2) | 1280 (46.8) | 3000 (75.2) | 4900 (28.2)

9. Secondary Outcome: AUC0-tau
Description: area under the curve over a dosing interval (tau)
Time Frame: as for outcome 3
Population: The pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of AM1476
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part B, Group 1: AM1476 100 mg QD | Part B, Group 2: AM1476 375 mg BID | Part B, Group 3: AM1476 500 mg BID
Number analyzed (Participants) | 6 | 6 | 6
h*ng/mL
  Day 1 | 77.7 (36.8) | 324 (43.6) | 702 (22.7)
  Day 10 | 110 (16.5) | 574 (30.6) | 953 (28.6)

10. Secondary Outcome: CL/F
Description: apparent total clearance
Time Frame: From pre-dose to up to 48 hours post-dose
Population: The pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of AM1476. At the 1 mg AM1476 dose level, the apparent total clearance was not calculable due to the limited quantifiable AM1476 concentrations available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Part A, Group 1: AM1476 1 mg | Part A, Group 2: AM1476 5 mg | Part A, Group 3: AM1476 25 mg | Part A, Group 4: AM1476 125 mg | Part A, Group 5: AM1476 375 mg | Part A, Group 6: AM1476 650 mg | Part A, Group 7: AM1476 950 mg | Part A, Group 8: AM1476 1500 mg | Part A, Group 9: AM1476 2400 mg
Number analyzed (Participants) | 0 | 5 | 6 | 6 | 6 | 6 | 5 | 6 | 6
L/h |  | 1480 (23.7) | 1550 (27.4) | 1080 (31.9) | 1030 (30.2) | 724 (71.8) | 620 (16.9) | 495 (75.0) | 487 (28.0)

11. Secondary Outcome: CL/F
Description: apparent total clearance
Time Frame: as for outcome 3
Population: The pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of AM1476
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Part B, Group 1: AM1476 100 mg QD | Part B, Group 2: AM1476 375 mg BID | Part B, Group 3: AM1476 500 mg BID
Number analyzed (Participants) | 6 | 6 | 6
L/h
  Day 1 | 1220 (35.0) | 1080 (45.6) | 673 (21.6)
  Day 10 | 906 (16.5) | 653 (30.6) | 525 (28.6)

12. Secondary Outcome: Vz/F
Description: apparent volume of distribution during the terminal phase
Time Frame: From pre-dose to up to 48 hours post-dose
Population: The pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of AM1476. At the 1 mg AM1476 dose level, the apparent volume of distribution during the terminal phase was not calculable due to the limited quantifiable AM1476 concentrations available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Part A, Group 1: AM1476 1 mg | Part A, Group 2: AM1476 5 mg | Part A, Group 3: AM1476 25 mg | Part A, Group 4: AM1476 125 mg | Part A, Group 5: AM1476 375 mg | Part A, Group 6: AM1476 650 mg | Part A, Group 7: AM1476 950 mg | Part A, Group 8: AM1476 1500 mg | Part A, Group 9: AM1476 2400 mg
Number analyzed (Participants) | 0 | 5 | 6 | 6 | 6 | 6 | 5 | 6 | 6
L |  | 5380 (35.6) | 10200 (30.8) | 13000 (60.7) | 20400 (163.0) | 10500 (92.7) | 7010 (13.0) | 6360 (75.5) | 5180 (43.2)

13. Secondary Outcome: Vz/F
Description: apparent volume of distribution during the terminal phase
Time Frame: as for outcome 3
Population: The pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of AM1476.
  A reliable characterization of the apparent volume of distribution during the terminal phase could not be obtained according the calculation criteria in the Statistical analytical plan for 2 participants dosed with 100 mg QD and 1 participant dosed with 375 mg BID on Day 10.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Part B, Group 1: AM1476 100 mg QD | Part B, Group 2: AM1476 375 mg BID | Part B, Group 3: AM1476 500 mg BID
Number analyzed (Participants) | 6 | 6 | 6
L
  Day 1 | 10100 (40.4) | 5020 (38.3) | 2800 (27.5)
  Day 10: number analyzed (Participants) | 4 | 5 | 6
  Day 10 | 14200 (29.4) | 12800 (37.0) | 12000 (48.9)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 7 weeks
Arm/Group | Part A, Groups 1 to 9: Placebo | Part A, Group 1: AM1476 1 mg | Part A, Group 2: AM1476 5 mg | Part A, Group 3: AM1476 25 mg | Part A, Group 4: AM1476 125 mg | Part A, Group 5: AM1476 375 mg | Part A, Group 6: AM1476 650 mg | Part A, Group 7: AM1476 950 mg | Part A, Group 8: AM1476 1500 mg | Part A, Group 9: AM1476 2400 mg | Part B, Groups 1 to 3: Placebo | Part B, Group 1: AM1476 100 mg QD | Part B, Group 2: AM1476 375 mg BID | Part B, Group 3: AM1476 500 mg BID
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/18 | 0/6 | 0/6 | 4/6 | 1/6 | 2/7 | 3/6 | 2/6 | 4/6 | 5/6 | 6/6 | 3/6 | 2/6 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A, Groups 1 to 9: Placebo (N=18) | Part A, Group 1: AM1476 1 mg (N=6) | Part A, Group 2: AM1476 5 mg (N=6) | Part A, Group 3: AM1476 25 mg (N=6) | Part A, Group 4: AM1476 125 mg (N=6) | Part A, Group 5: AM1476 375 mg (N=7) | Part A, Group 6: AM1476 650 mg (N=6) | Part A, Group 7: AM1476 950 mg (N=6) | Part A, Group 8: AM1476 1500 mg (N=6) | Part A, Group 9: AM1476 2400 mg (N=6) | Part B, Groups 1 to 3: Placebo (N=6) | Part B, Group 1: AM1476 100 mg QD (N=6) | Part B, Group 2: AM1476 375 mg BID (N=6) | Part B, Group 3: AM1476 500 mg BID (N=6)
Palpitations (Cardiac disorders) | 0 | NA | NA | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ocular discomfort (Eye disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | NA | NA | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | NA | NA | 0 | 0 | 0 | 2 | 1 | 4 | 3 | 0 | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | NA | NA | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Application site erythema (General disorders) | 1 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site rash (General disorders) | 0 | NA | NA | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site erythema (General disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Chest pain (General disorders) | 0 | NA | NA | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | NA | NA | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | NA | NA | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | NA | NA | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | NA | NA | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | NA | NA | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | NA | NA | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1
Dizziness Postural (Nervous system disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | NA | NA | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 1
Lethargy (Nervous system disorders) | 0 | NA | NA | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | NA | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/15/NCT04691115/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT04691115/SAP_001.pdf